CLINICAL TRIAL: NCT05536544
Title: The Inflammatory Bowel Disease Mediterranean Diet (IBDMED) Microbiome-targeting Nutritional Education Program for CD Control and Prevention
Brief Title: The Inflammatory Bowel Disease Mediterranean Diet (IBDMED) Microbiome-targeting Nutritional Education Program
Acronym: IBDMED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Asian Institute of Gastroenterology (Unknown)
Responsible Party: Principal Investigator, IRIS DOTAN, Head of The Gastroenterology Division, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 0359-21
Record Dates: First submitted 2022-09-01; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Inflammatory Bowel Diseases
Keywords: IBD
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBDMED-ISR (Other): Patients with newly diagnosed CD in Israel
  Interventions: Other: IBDMED; Other: Control
- IBDMED-IND (Other): Patients with newly diagnosed CD in India
  Interventions: Other: IBDMED; Other: Control

INTERVENTIONS:
Other: IBDMED — The IBDMED program will be applied for 8 weeks and include education on MED diet and lifestyle components, focused on increasing and diversifying dietary fiber intake, reduction of ultra-processed food intake and promoting an active lifestyle. This intervention is digitally supported by an interactive website application and step trackers to monitor lifestyle parameters.
Other: Control — Dietary counseling according to the local dietary guidelines for patients with IBD

SUMMARY:
The rising incidence of Crohn's disease (CD) and ulcerative colitis (UC), especially in the newly industrialized nations of Asia, highlights the possible role of environmental triggers such as diet and the gut microbiome in the pathogenesis of inflammatory bowel diseases (IBD). The Mediterranean diet (MED) has been previously correlated with beneficial outcomes in several chronic and immune-mediated diseases and has been linked with positive outcomes in IBD. However, consumption of high fiber foods like fruits, vegetables, whole grains, legumes and nuts may be challenging for patients with IBD without tight dietary guidance and support.

The IBDMED nutritional education program aims to improve the adherence of patients with IBD to MED. Patients are educated on how to implement and incorporate MED principles into their daily lifestyle, by providing information, tips, practical tools, cooking methods and recipes, that are available on an interactive website and application. Patients are monitored for their diet, sleep, physical activity and stress levels via fitness trackers and questionnaires developed for this study and receive feedback and personal recommendations from the study dietitians along the way.

This RCT will assess the feasibility and effects of an 8-week IBDMED nutritional and lifestyle education program vs. the nutritional standard of care in patients with newly diagnosed CD and in healthy subjects in Israel and India.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with early CD, defined as up to 12 months from diagnosis
2. Inflammatory (B1) phenotype, specifically-no known fibrostenotic (B2) or internal penetrating (B3) disease. No known perianal disease (p). Any CD location will be included (L1-4)
3. Patients with mild CD as measured by HBI 5-7 or CDAI 150-220 or patients with HBI<5 or CDAI<150 with at least one additional objective measure of inflammation: 1. inflammatory biomarkers: elevated CRP or fecal calprotectin at enrollment; active disease by endoscopy or VCE performed up to 12 weeks prior to enrollment; active inflammation demonstrated by imaging (CTE, MRE, IUS) performed up to 12 weeks prior to enrollment.
4. Any stable concomitant CD therapy is allowed. 5-ASA (stable dose for at least 2 weeks), steroids (budesonide or any non topical corticosteroids)-stable dose for at least 2 weeks: prednisone up to 20 mg/day or budesonide up to 6 mg/day; immunomodulators (stable dose for 8 weeks) and/ or anti-TNFs at least 4 weeks after the end of induction or any optimization; anti integrins at least 4 weeks after the end of induction or any optimization; anti IL12/IL23 at least 4 weeks after the end of induction or any optimization; None of the above. For inclusion in a non-steroid group, a 2-week washout period will be required.
5. TB evaluation was done in the Indian population
6. For India-Hindi/Telugu speakers
7. Willing and able to sign an informed consent form
8. Willing and able to participate and adhere to IBDMED program

Exclusion Criteria:

1. Pregnant women
2. Diabetes mellitus
3. Any previous gastrointestinal surgery (except appendectomy)
4. Antibiotic therapy during the 4 weeks prior to enrollment. After enrollment, a non-CD short course of antibiotics will be allowed, if prescribed
5. Any concomitant disease or treatment that according to the treating physician considerations interferes with patient safety or study outcomes (specifically-uncontrolled thyroid disease, renal failure)
6. Undernutrition or need for enteral nutrition supplementation according to the treating dietitian

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Composite biological score | 8 weeks
  A composite biological score comprised of changes in clinical (HBI/CDAI), inflammatory (CRP/calprotectin) and microbial (diversity, MDI) indices. A decrease in clinical indices, inflammatory markers or MDI will be considered positive and will be scored as follows: -10%: +1 point, -20%: +2 points, -30%: +3 points; An increase in microbial diversity will be considered positive and will be scored as follows: +10%: +1 point, +20%: +2 points, +30%: +3 points. The composite biological score ranges between 0-15 points.

SECONDARY OUTCOMES:
Clinical and inflammatory response | 8 weeks
  Decrease in inflammatory activity: at least 30% decrease in HBI and/or CDAI and the additional inflammatory biomarker used at inclusion. In any case where CRP or fecal calprotectin were elevated, they will be used to evaluate decreased activity.
Improvement in quality of life | 8 weeks
  Improved quality of life as assessed by the PRO2 (≥50% or ≥ 4 points)
Dietary adherance | 8 weeks
  Adherence to IBDMED in India and Israel-measured by IBDMED score. The IBDMED adherance screener includes 11 items and ranges between 0-30.

OTHER OUTCOMES:
Microbial outcomes- alpha diversity | 8 weeks
  Microbial diversity will be compared between groups and intra-individual changes will be assessed using paired analysis.
Microbial outcomes- Microbial dysbiosis index | 8 weeks
  MDI will be compared between groups and intra-individual changes will be assessed using paired analysis.

CONTACTS AND LOCATIONS:
Locations (2):
- Asian Institute of Gastroenterology, Hyderabad, India
- Rabin Medical Center, Petah Tikva, Israel